CLINICAL TRIAL: NCT04852679
Title: A Phase 3, Single-arm, Open-label, Multicentre Study to Assess the Efficacy and Safety of Deep Subcutaneous Injections of Lanreotide Autogel® 120 mg Administered Every 28 Days in Chinese Participants With Unresectable, Locally Advanced or Metastatic Grade 1 or 2 Gastroenteropancreatic Neuroendocrine Tumours (GEP-NETs)
Brief Title: Study to Assess the Efficacy and Safety of Lanreotide Autogel® in Chinese Participants With GEP-NETs
Acronym: PALACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-CN-52030-411
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lanreotide Autogel 120 mg (Other): Subjects will be treated with lanreotide Autogel® 120mg, every 28 days (+/- 3 days).
  Interventions: Drug: Lanreotide autogel

INTERVENTIONS:
Drug: Lanreotide autogel — Administered as deep subcutaneous (SC) injections

SUMMARY:
This study will be conducted to support the registration of the lanreotide Autogel 120 mg formulation in China for the treatment of GEP-NETs and treatment of clinical symptoms of NETs.

The study will include a screening period of up to 4 weeks followed by a 48-week intervention period. After completion of the main study period, five participants will continue in a self/partner injection cohort with lanreotide Autogel 120 mg every 28 days for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Male or female of 18 years of age or older when informed consent is obtained
* Has a histologically proven Grade 1 or 2 GEP-NET according to WHO (World Health Organisation) classification
* Has an unresectable metastatic or locally advanced NET.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status lower or equal to 2.

Exclusion Criteria:

* Participants with poorly differentiated Gastroenteropancreatic neuroendocrine carcinoma (GEP-NEC), high-grade GEP-NEC and goblet cell carcinoid.
* Has been treated with octreotide acetate long-acting release or lanreotide acetate Autogel formulation within 8 weeks prior to screening tests or lanreotide PR 40 mg within 4 weeks prior to screening tests.
* Has been treated with subcutaneous or intravenous octreotide acetate within 1 week prior to screening tests.
* Has been treated with mammalian target of rapamycin (mTOR) inhibitors or multi-target tyrosine kinase (MTK) inhibitors within 4 weeks prior to screening tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (14):
- China (14):
  - Cancer Hospital Chinese Academy of Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Qilu Hospital Of Shandong University, Jinan, Shandong
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Centre, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The second affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Where patient data can be anonymised, Ipsen will share all individual participant data that underlie the results reported in the published journal article with qualified researchers who provide a valid research question. Study documents, such as the study protocol and clinical study report, are not always available.
Time Frame: Data are available beginning 6 months and ending 5 years after the publication of the findings in a journal; after this time, only raw data may be available.
Access Criteria: Proposals should be submitted to DataSharing@ipsen.com and will be assessed by a scientific review board.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3 single-arm, open-label study was conducted in chinese adult participants with unresectable, locally advanced or metastatic Grade 1 or 2 gastroenteropancreatic neuroendocrine tumours (GEP-NETs) at 14 investigational sites in China between 24 May 2021 and 13 January 2023.
Pre-assignment Details: This study consisted of a screening period (up to 4 weeks), followed by a 48-week main intervention period and then a 24-week independent injection period. A total of 43 participants were treated in this study.
Groups:
- Lanreotide Autogel 120 Milligram (mg): All participants received a fixed dose of lanreotide autogel 120 mg subcutaneous (SC) injection every 28 days up to 48 weeks during the main intervention period. After completion of the main intervention period, eligible participants entered an independent injection period to receive lanreotide autogel 120 mg SC injection every 28 days for 24 weeks.
Period: Main Intervention Period
Arm/Group | Lanreotide Autogel 120 Milligram (mg)
Started (Treated participants.) | 43
Study Intervention Completion at Week 24 | 28
Completed (Study intervention completion at Week 48.) | 22
Not Completed | 21
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 16
Not completed — Refused study visit | 1
Period: Independent Injection Period
Arm/Group | Lanreotide Autogel 120 Milligram (mg)
Started | 5 (Only eligible participants were rolled over to independent injection period.)
Completed (Study intervention completion at Week 72.) | 4
Not Completed | 1
Not completed — Missed study visit | 1

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) analysis set included all participants who received at least 1 dose of study intervention.
Groups:
- Lanreotide Autogel 120 mg: All participants received a fixed dose of lanreotide autogel 120 mg SC injection every 28 days up to 48 weeks during the main intervention period. After completion of the main intervention period, eligible participants entered an independent injection period to receive lanreotide autogel 120 mg SC injection every 28 days for 24 weeks.
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 43
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) of Tumour Response Assessed by Blinded Independent Central Review (BICR) at Week 24
Description: The CBR was defined as the percentage of participants with a best overall response of confirmed complete response (CR), confirmed partial response (PR), or continued stable disease (SD) until the time of assessment according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria v1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 24
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
percentage of participants | 62.79 [46.7 to 77.0]

2. Secondary Outcome: Progression Free Survival (PFS) by BICR Within Weeks 24 and 48
Description: The PFS was defined as the time from the first administration of study intervention to the date of the first documented PD measured using RECIST criteria v1.1 and confirmed by BICR, or death from any cause, whichever comes first. The PFS was estimated using the Kaplan-Meier method. The PD was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 24 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
weeks
  Week 24 | NA [24.1 to NA] — Medium and upper limit of confidence interval (CI) could not be determined as too few survival events during the 24 weeks study duration.
  Week 48 | NA [36.1 to NA] — Medium and upper limit of CI could not be determined as too few survival events during the main intervention period.

3. Secondary Outcome: Overall Survival (OS) at the End of the Main Intervention Period
Description: The OS was defined as the time from the first administration of study intervention to the date of death from any cause. The OS was estimated using the Kaplan-Meier method.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Week 48 (end of the main intervention period)
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
weeks | NA [NA to NA] — The results could not be determined as too few death events during the main intervention period.

4. Secondary Outcome: Time to Progression (TTP) During Main Intervention Period
Description: The TTP was defined as the time from the first administration of study intervention to the date of the first documented PD, or clinical progression confirmed by the investigator. The TTP was assessed by BICR and estimated using the Kaplan-Meier method. The PD was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 12, 24, 36 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
weeks | NA [48.0 to NA] — Medium and upper limit of CI could not be determined as too few progression events during the main intervention period.

5. Secondary Outcome: Percentage of Participants Alive and Without Tumour Progressive at Weeks 24 and 48
Description: Percentage of participants who were alive and progression free per RECIST v1.1 using BICR assessments at 24 and 48 weeks after first dose of study intervention were reported. The PFS was estimated using the Kaplan-Meier method. The PD was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 24 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
percentage of participants
  Week 24 | 77.4 [59.6 to 88.1]
  Week 48 | 59.0 [36.1 to 76.1]

6. Secondary Outcome: Clinical Benefit Rate Assessed by BICR at Week 48
Description: The CBR was defined as the percentage of participants with a best overall response of confirmed CR, confirmed PR, or continued SD until the time of assessment according to RECIST criteria v1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Week 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
percentage of participants | 58.1 [42.1 to 73.0]

7. Secondary Outcome: Overall Response Rate (ORR) at Weeks 24 and 48
Description: The ORR was defined as the percentage of participants with a best overall response of confirmed CR or confirmed PR. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 24 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
percentage of participants
  Week 24 | 0 [0.0 to 8.2]
  Week 48 | 7.0 [1.5 to 19.1]

8. Secondary Outcome: Disease Control Rate (DCR) at Weeks 24 and 48
Description: The DCR was defined as the percentage of participants with a best overall response of confirmed CR, confirmed PR or SD. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study intervention) and Weeks 24 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
percentage of participants
  Week 24 | 69.8 [53.9 to 82.8]
  Week 48 | 69.8 [53.9 to 82.8]

9. Secondary Outcome: Number of Participants With Neuroendocrine Tumours (NET)-Related Clinical Symptoms at Weeks 24 and 48
Description: The presence or absence of endocrine symptoms of NETs (example; flushing, diarrhoea, abdominal pain, weakness, heartburn, nausea, vomiting, sweating, tremor, palpitation, or erythema) were assessed by the investigator at screening. In participants with symptoms of NETs at screening, a baseline assessment of the symptoms experienced in the last 4 weeks was performed by questioning before study intervention administration at Day 1. These symptoms were recorded in the case report form and severity graded upon National Cancer Institute Common Terminology Criteria for Adverse Events. Where, Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death.
Time Frame: Weeks 24 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 43
Participants
  Week 24: Diarrhea: Grade 1 | 0
  Week 24: Diarrhea: Grade 2 | 0
  Week 24: Diarrhea: Grade 3 | 0
  Week 24: Diarrhea: Grade 4 | 0
  Week 24: Diarrhea: Grade 5 | 0
  Week 24: Diarrhea: Missing | 43
  Week 48: Diarrhea: Grade 1 | 0
  Week 48: Diarrhea: Grade 2 | 0
  Week 48: Diarrhea: Grade 3 | 0
  Week 48: Diarrhea: Grade 4 | 0
  Week 48: Diarrhea: Grade 5 | 0
  Week 48: Diarrhea: Missing | 43
  Week 24: Hypertension: Grade 1 | 1
  Week 24: Hypertension: Grade 2 | 0
  Week 24: Hypertension: Grade 3 | 0
  Week 24: Hypertension: Grade 4 | 0
  Week 24: Hypertension: Grade 5 | 0
  Week 24: Hypertension: Missing | 42
  Week 48: Hypertension: Grade 1 | 0
  Week 48: Hypertension: Grade 2 | 0
  Week 48: Hypertension: Grade 3 | 0
  Week 48: Hypertension: Grade 4 | 0
  Week 48: Hypertension: Grade 5 | 0
  Week 48: Hypertension: Missing | 43
  Week 24: Nodal tachycardia: Grade 1 | 0
  Week 24: Nodal tachycardia: Grade 2 | 0
  Week 24: Nodal tachycardia: Grade 3 | 0
  Week 24: Nodal tachycardia: Grade 4 | 0
  Week 24: Nodal tachycardia: Grade 5 | 0
  Week 24: Nodal tachycardia: Missing | 43
  Week 48: Nodal tachycardia: Grade 1 | 0
  Week 48: Nodal tachycardia: Grade 2 | 0
  Week 48: Nodal tachycardia: Grade 3 | 0
  Week 48: Nodal tachycardia: Grade 4 | 0
  Week 48: Nodal tachycardia: Grade 5 | 0
  Week 48: Nodal tachycardia: Missing | 43

10. Secondary Outcome: Change From Baseline in Plasma Chromogranin A (CgA) at Weeks 12, 24, 36 and 48
Description: The CgA determination was useful for staging, prognosis and follow up, since the serum concentration correlated to the tumour mass. Blood samples were collected to measure circulating CgA.
Time Frame: Baseline (within 28 days before start of study intervention) and Weeks 12, 24, 36 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: microgram per liter
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
microgram per liter
  Week 12 | -35.7305 (105.1477)
  Week 24: number analyzed (Participants) | 25
  Week 24 | -46.2278 (126.1348)
  Week 36: number analyzed (Participants) | 24
  Week 36 | -51.8435 (125.4386)
  Week 48: number analyzed (Participants) | 19
  Week 48 | -30.8557 (134.5523)

11. Secondary Outcome: Change From Baseline in 5-Hydroxyindoleacetic Acid (5-HIAA) at Weeks 12, 24, 36 and 48
Description: Urine samples were collected to measure 5-HIAA.
Time Frame: Baseline (within 28 days before start of study intervention) and Weeks 12, 24, 36 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: milligram per liter
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
milligram per liter
  Week 12 | -0.5495 (0.9598)
  Week 24: number analyzed (Participants) | 25
  Week 24 | -1.1965 (4.5374)
  Week 36: number analyzed (Participants) | 23
  Week 36 | -0.0837 (1.6261)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -1.3129 (6.3055)

12. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Assessment at Weeks 12, 24, 36 and 48
Description: The European Organization for Research and Treatment of Cancer QoL Questionnaire for Cancer participants contains 30 single items. For questions 1 to 28, score ranges from 1 to 4 where, 1= not at all, 2= a little, 3= quite a bit and 4= very much. Global health status/QoL contains questions 29 and 30 and score ranges from 1 to 7, where 1= very poor and 7= excellent. Total score ranges from 0 (poor) to 100 (excellent). Higher score indicates a high QoL.
Time Frame: Baseline (within 28 days before start of study intervention) and Weeks 12, 24, 36 and 48
Population: The ITT analysis set included all participants who received at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lanreotide Autogel 120 mg
Number analyzed (Participants) | 36
units on a scale
  Week 12 | 3.0 (16.0)
  Week 24: number analyzed (Participants) | 25
  Week 24 | -4.0 (18.2)
  Week 36: number analyzed (Participants) | 24
  Week 36 | -9.4 (16.5)
  Week 48: number analyzed (Participants) | 20
  Week 48 | -13.8 (19.0)

ADVERSE EVENTS:
Time Frame: Main intervention period: Treatment-emergent adverse events (TEAEs) were reported from first injection of study intervention up to Week 48, approximately 48 weeks. Independent injection period: TEAEs were reported from Week 48 to end of study or 4 weeks after last injection of study intervention, approximately 28 weeks.
Description: Main intervention period: The safety set included all participants who received at least 1 dose of study intervention.
  Independent injection period: The independent injection set included all participants who received the study intervention by independent injection.
  A TEAE is defined as any adverse event that is not occurred prior to the first dose of study intervention or occurred prior to the first dose of study intervention but the intensity increased during the active phase of the study.
Groups:
- Main Intervention Period: Lanreotide Autogel 120 mg: All participants received a fixed dose of lanreotide autogel 120 mg SC injection every 28 days up to 48 weeks.
- Independent Injection Period: Lanreotide Autogel 120 mg: Eligible participants received a fixed dose of lanreotide autogel 120 mg SC injection every 28 days for 24 weeks.
Arm/Group | Main Intervention Period: Lanreotide Autogel 120 mg | Independent Injection Period: Lanreotide Autogel 120 mg
All-Cause Mortality (participants affected / at risk) | 2/43 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/43 | 0/5
Other Adverse Events (participants affected / at risk) | 43/43 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Intervention Period: Lanreotide Autogel 120 mg (N=43) | Independent Injection Period: Lanreotide Autogel 120 mg (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Intervention Period: Lanreotide Autogel 120 mg (N=43) | Independent Injection Period: Lanreotide Autogel 120 mg (N=5)
Alanine aminotransferase increased (Investigations) | 9 (10) | 0 (0)
Bilirubin conjugated increased (Investigations) | 8 (8) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (9) | 0 (0)
Weight decreased (Investigations) | 8 (10) | 0 (0)
Blood glucose increased (Investigations) | 7 (7) | 0 (0)
White blood cell count decreased (Investigations) | 6 (8) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 5 (5) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 4 (4) | 0 (0)
Weight increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Blood urea increased (Investigations) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
Red blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 18 (32) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (8) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (8) | 0 (0)
Injection site nodule (General disorders) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT04852679/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT04852679/SAP_001.pdf